CLINICAL TRIAL: NCT02825394
Title: Specific Point-of-Care Testing of Coagulation in Patients Treated With Direct Oral Anticoagulants Part 1
Brief Title: Specific PoC Testing of Coagulation in Patients Treated With DOAC 1
Acronym: SPOCT-DOAC 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other)
Responsible Party: Principal Investigator, Dr. Sven Poli, MD MSc, University Hospital Tuebingen
Other Study IDs: 270/2015BO1
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Anticoagulation With NOAC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples, citrated blood samples and citrated plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- apixaban initiation: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)
- apixaban on-treatment: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)
- dabigatran initiation: N=20
  Interventions: Other: ecarin clotting time point-of-care testing (ECT-POCT)
- dabigatran on-treatment: N=20
  Interventions: Other: ecarin clotting time point-of-care testing (ECT-POCT)
- rivaroxaban initiation: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)
- rivaroxaban on-treatment: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)
- edoxaban initiation: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)
- edoxaban on-treatment: N=20
  Interventions: Other: anti-Xa activity point-of-care testing (aXa-POCT)

INTERVENTIONS:
Other: anti-Xa activity point-of-care testing (aXa-POCT)
  Other Names: Cascade Abrazo with ENOX and ENOX LR test cards
  Groups: apixaban initiation; apixaban on-treatment; edoxaban initiation; edoxaban on-treatment; rivaroxaban initiation; rivaroxaban on-treatment
Other: ecarin clotting time point-of-care testing (ECT-POCT)
  Other Names: Cascade Abrazo with DTM test cards
  Groups: dabigatran initiation; dabigatran on-treatment

SUMMARY:
The investigators study aims to test the correlation between the Cascade Abrazo point-of-care testing (POCT) device (Helena Laboratories, USA) and plasma levels of apixaban, dabigatran, edoxaban and rivaroxaban, and to determine the diagnostic accuracy of POCT to rule out or detect relevant levels of direct oral anticoagulants (DOAC) in real-life patients.

ELIGIBILITY:
Inclusion Criteria:

* Part A only: planned initiation of treatment with apixaban, dabigatran, edoxaban or rivaroxaban
* Part B only: ongoing treatment with apixaban, dabigatran, edoxaban or rivaroxaban
* Age ≥ 18 years
* Written informed consent by patient

Exclusion Criteria:

* Part A only: intake of vitamin K antagonists or direct oral anticoagulants (DOAC) ≤ 14 days prior to study participation
* Part B only: intake of vitamin K antagonists or different DOAC ≤ 14 days prior to study participation
* Intake of unfractionated heparin ≤ 12 hours, low-molecular-weight heparin ≤ 24h, heparinoids (e.g. fondaparinux) ≤ 72h, or direct thrombin inhibitors other than dabigatran ≤ 72h prior to study participation
* Part A only: abnormal routine coagulation test values at baseline (defined by INR > 1.2, Quick < 70% or aPTT > 40 sec)
* History of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Part A: patients, who are newly started on oral anticoagulation with apixaban, dabigatran, edoxaban or rivaroxaban for secondary prevention of thromboembolic events.
  Part B: patients, on-treatment with apixaban, dabigatran, edoxaban or rivaroxaban.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-10-13 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of direct oral anticoagulant (DOAC) plasma concentration with Cascade Abrazo point-of-care testing (POCT) result | 24 hours
  DOAC concentrations determined by ultra-performance liquid chromatography-tandem mass spectrometry

SECONDARY OUTCOMES:
Diagnostic accuracy (sensitivity and specificity) of the Cascade Abrazo POCT to rule out or detect relevant DOAC plasma levels | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based prothrombin time (PT) assay | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based activated thromboplastin time (aPTT) assay | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based thrombin time (TT) assay | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based diluted thrombin time (dTT) assay | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based ecarin clotting time (ECT) assay | 24 hours
Correlation of DOAC plasma concentrations with laboratory-based anti-Xa activity assay | 24 hours
Correlation of edoxaban plasma concentrations with CoaguChek point-of-care prothrombin time (PT) assay | 24 hours
Correlation of edoxaban plasma concentrations with Hemochron Signature point-of-care prothrombin time (PT) assay | 24 hours
Correlation of edoxaban plasma concentrations with Hemochron Signature point-of-care activated thromboplastin time (aPTT) assay | 24 hours
Correlation of edoxaban plasma concentrations with Hemochron Signature point-of-care activated clotting time plus (ACT+) assay | 24 hours
Correlation of edoxaban plasma concentrations with Hemochron Signature point-of-care activated clotting time low-range (ACT-LR) assay | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hartig F, Birschmann I, Peter A, Horber S, Ebner M, Sonnleitner M, Spencer C, Bombach P, Stefanou MI, Tunnerhoff J, Mengel A, Kuhn J, Ziemann U, Poli S. Point-of-care testing for emergency assessment of coagulation in patients treated with direct oral anticoagulants including edoxaban. Neurol Res Pract. 2021 Mar 1;3(1):9. doi: 10.1186/s42466-021-00105-4. PMID 33641678
- [Derived] Hartig F, Birschmann I, Peter A, Ebner M, Spencer C, Gramlich M, Richter H, Kuhn J, Lehmann R, Blumenstock G, Zuern CS, Ziemann U, Poli S. Specific Point-of-Care Testing of Coagulation in Patients Treated with Dabigatran. Thromb Haemost. 2021 Jun;121(6):782-791. doi: 10.1055/s-0040-1721775. Epub 2021 Jan 14. PMID 33469905